CLINICAL TRIAL: NCT00374998
Title: A Phase I Study to Assess the Safety and Immunogenicity of the Polyprotein Malaria Vaccine Candidates FP9 PP and MVA PP in Healthy Adults Using a Prime-Boost Delivery Schedule
Brief Title: Safety and Immunogenicity Study of the Malaria Vaccines FP9 PP and MVA PP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Vaccine Initiative (Other)
Collaborators: University of Oxford (Other); Wellcome Trust (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC027.1; EudraCT number: 2004-002424-17; EMVI trial identifier: PP_1_04
Record Dates: First submitted 2006-09-10; First posted 2006-09-12 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Malaria, Falciparum; Malaria
Keywords: Malaria; Vaccine; Prime-boost
MeSH Terms: conditions — Malaria, Falciparum; Malaria

INTERVENTIONS:
Biological: FP9-PP (FP9 polyprotein)
Biological: MVA-PP (Modified Virus Ankara polyprotein)

SUMMARY:
This study examines two new malaria vaccines (FP9-PP and MVA-PP) in healthy human volunteers to determine their safety and ability to induce a measurable immune response against malaria.

DETAILED DESCRIPTION:
Malaria infection kills over 2 million people each year. It is a major problem for those who live in endemic areas and for travellers. There is clearly a great need for a safe effective malaria vaccine.

The purpose of this study is to test two candidate malaria vaccines (FP9-PP and MVA-PP) in different concentrations and combinations. These live viral vectors encode a 'polyprotein' of six fused malaria antigens expressed at liver and blood stages of the malaria parasite lifecycle. MVA-PP uses the Modified Virus Ankara vector, a weakened form of the smallpox vaccine, vaccinia. FP9-PP uses a highly attenuated avian pox virus (FP9) as the vector instead. The two vaccines will be used in combination in a 'prime boost' strategy to enhance the response of the cellular immune system.

This study will:

1. Examine safety
2. Examine immunogenicity
3. Provide a subgroup of vaccinated volunteers to test clinical efficacy in the following malaria challenge study (VAC027.2)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Resident in or near Oxford, UK for the duration of the vaccination study
* Willingness to allow the investigators to access hospital and General Practitioner medical notes
* For females only, willingness to practice continuous effective contraception during the study and if participating, during the subsequent challenge study.
* Agreement to refrain from blood donation during the course of the study
* Written informed consent
* Willingness to undergo an HIV test

Exclusion Criteria:

* Any deviation from the protocol-defined normal range in biochemistry or haematology blood tests or in urine analysis
* Prior receipt of an investigational malaria vaccine
* Use of any investigational or non-registered drug, vaccine or medical device other than the study vaccine within 30 days preceding dosing of study vaccine, or planned use during the study period
* Administration of chronic immunosuppressive drugs or other immune modifying drugs within six months of vaccination
* History of malaria chemoprophylaxis with chloroquine within 5 months prior to the planned challenge, with Lariam within 6 weeks prior to the challenge, and Riamet within 2 weeks prior to the challenge
* Any history of malaria
* Travel to a malaria endemic country within the previous 6 months prior to the planned challenge
* Planned travel to malarious areas during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection and asplenia
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products
* Evidence of cardiovascular disease
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of haemoglobinopathies
* History of diabetes mellitus
* Chronic or active neurological disease
* Chronic gastrointestinal disease
* History of more than 2 hospitalisations for invasive bacterial infections
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* Evidence of serious psychiatric condition
* Any other on-going chronic illness requiring hospital specialist supervision

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35
Dates: Start 2006-04; Study Completion 2007-01

PRIMARY OUTCOMES:
Immediate reactogenicity
Adverse events occurring before the end of the trial
Biological safety (haematological and biochemical indices)

SECONDARY OUTCOMES:
T-cell immunogenicity (prime-boost groups)
Humoral immunogenicity (prime-boost groups)
Gene expression (prime-boost groups)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian VS Hill, MA, BM BCh, DPhil, DM, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology & Tropical Medicine, University of Oxford, Oxford, United Kingdom